CLINICAL TRIAL: NCT07333820
Title: Clinical Study to Evaluate the Safety and Anti-Tumor Activity of AB-201 in Subjects With Advanced HER2 Positive Gastric/Gastroesophageal Junction(GEJ) Cancer
Brief Title: Clinical Study to Evaluate the Safety and Anti-Tumor Activity of AB-201
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4-2025-0975
Record Dates: First submitted 2025-12-15; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Malignant Neoplasm of Stomach, Unspecified
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AB-201 Dose escalation (Experimental): * Drug: AB-201
  * Drug: Cyclophosphamide
  * Drug: Fludarabine
  Interventions: Drug: AB-201 Dose escalation

INTERVENTIONS:
Drug: AB-201 Dose escalation — 1. Lymphodepletion Before administration of of AB-201, subjects will receive a lymphodepleting regimen consisting of cyclophosphamide (500 mg/m2/day IV) and fludarabine (30 mg/m2/day IV) to induce lymphocyte depletion and create an optimal environment for expansion of AB-201 in vivo.
     However, the lymphodepletion regimen may be adjusted according to the regulations of the institution or at the discretion of the principal investigator.
  2. AB-201 Administration A total of one dose of AB-201 (adjusted for a subject's body weight) as IV infusions are planned during the treatment phase.
  <Dose Levels for AB-201(adjusted for a subject's body weight)>
  1. Starting dose: 5.0 × 10^5 cells/kg
  2. 1.5 × 10^6 cells/kg
  3. 5.0 × 10^6 cells/kg

SUMMARY:
HER2 is highly expressed on the surface of several cancer types, including breast and gastric/gastroesophageal junction (GEJ) cancers. Several commercially available HER2-directed oncology therapies exist; however, most patients who initially derive meaningful clinical benefit from these agents eventually relapse or experience disease progression. Accordingly, the development of safe and effective treatments for patients who have exhausted current HER2-directed options remains an important unmet medical need.

AB-201 has demonstrated direct, HER2-specific, and potent cytotoxicity against multiple tumor cell lines both in vitro and in vivo. In addition, AB-201 has shown the ability to secrete cytokines, including tumor necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ), upon activation. Based on this emerging HER2-targeted cell therapy dataset, a HER2 CAR-NK therapy such as AB-201 may offer a safe, active, and readily available treatment option for patients with HER2-positive solid tumors.

This clinical trial will enroll subjects with HER2-positive gastric/GEJ cancers. The primary objective of the study is to evaluate the safety and tolerability of AB-201 in subjects with advanced HER2-positive gastric/GEJ cancers. The secondary objective is to assess the preliminary efficacy of AB-201, measured by objective response rate (ORR) per RECIST v1.1, in subjects with advanced gastric/GEJ cancers.

DETAILED DESCRIPTION:
Study designed to evaluate the safety, tolerability, and efficacy of AB-201 in subjects with advanced HER2 positive gastric/GEJ cancers.

Up to 18 subjects will be enrolled, and the study will be conducted by dose escalation.

During the Dose Escalation stage of this study, up to 3 escalating dose levels of AB-201 will be explored. The maximum tolerated dose (MTD) and/or maximum administered dose (MAD) for AB-201 will be defined as the highest dose level at which not more than 1 of 6 subjects in a cohort experiences a dose-limiting toxicity (DLT) as outlined below. The highest dose administered becomes the MAD if the MTD is not reached.

AB-201 is a cryopreserved, infusion-ready suspension cell therapy comprised of ex vivo-expanded allogeneic cord blood-derived NK cells that have been genetically modified to express a HER2-directed CAR and secrete IL-15.

AB-201 will be administered as a single IV infusion starting at 48 hours (but no more than 7 days) after completion of the lymphodepletion regimen. A 28-day observation period will then occur, at the end of which all relevant safety data will be reviewed.

Study participation for each subject begins with up to 28 days (1 month) of screening following written informed consent, then lymphodepletion treatment, followed by AB-201. All subjects will be monitored for a total duration of 18 months of follow-up from the administration of AB-201.

Safety will be assessed according to the Schedule of Activities by monitoring AEs (including DLTs, AEs of special interest [AESIs], and serious AEs [SAEs]), concomitant medications, physical examinations, ECOG performance status, acute GvHD, vital signs, and laboratory test findings. As an additional safety measure, Bayesian stopping bounds will be employed for the duration of the study.

Disease assessments will be performed according to the Schedule of Activities per RECIST v1.1. Imaging scans (CT or MRI) will be performed at Months 1, 2, 3, 6, 9, 12, 15, and 18 for efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Males or females ≥ 19 years of age at the time of informed consent.
3. The ECOG performance status 0 to 1.
4. Patients with an expected survival of at least 3 months
5. Histologically confirmed HER2-expressed gastric/GEJ cancer ≥IHC 1+ within 36 months prior to study entry.
6. Confirmed diagnosis (pathologically documented) of an advanced/unresectable or metastatic HER2+ gastric/GEJ cancer that is refractory to, or intolerable of standard treatment, or for which no standard treatment is available.
7. Prior cancer therapies per the National Comprehensive Cancer Network (NCCN) guidelines

   1. Subjects with gastric/GEJ cancer must have received ≥ 2 prior systemic therapy(ies)
   2. Subjects with IHC 3+ or IHC 2+/ISH+ cancers must have received previous treatment with a HER2-targeting therapy
   3. If the investigator determines no standard treatment remains
8. Has adequate treatment washout period prior receiving AB-201, defined as:

   * Major surgery ≥ 4 weeks
   * Radiation therapy ≥ 4 weeks (if palliative stereotactic radiation therapy without abdominal, ≥ 2 weeks)
   * Autologous transplantation ≥ 3 months
   * Chemotherapy (including antibody-drug therapy) ≥ 3 weeks (≥ 2 weeks for 5-fluorouracil-based agents, folinate agents and/or weekly paclitaxel. ≥ 6 weeks for nitrosoureas or mitomycin C, > 1 week for TKIs approved for the treatment of breast or gastric/GEJ cancers - baseline computed tomography (CT) scan must be completed after discontinuation of TKI)
   * Hormonal therapy ≥ 3 weeks
   * Immunotherapy ≥ 4 weeks
9. Measurable disease or non-measurable but evaluable disease according to RECIST v1.1, as assessed by computed tomography (CT) or magnetic resonance imaging (MRI), with at least one measurable or non-measurable but evaluable lesion.
10. Oxygen saturation via pulse oximeter ≥ 92% at rest on room air
11. Left ventricular ejection fraction (LVEF) ≥ 50% and no evidence of pericardial effusion as determined by an echocardiogram (ECHO)/multigated acquisition (MUGA) scan
12. Baseline laboratory values fulfilling the following requirements to demonstrate adequate hematologic, renal, and hepatic function:

    * Absolute neutrophil count (ANC) ≥ 1000/mm3 (1.0 × 109/L)
    * Platelets (PLT) ≥ 75000/mm3 (75 × 109/L)
    * Hemoglobin ≥ 8.0 g/dL (transfusions are allowed up to 2 weeks prior to the first AB-201 dose and, as needed, during the treatment period.)
    * Creatinine clearance ≥ 45 mL/min using the Cockcroft-Gault equation, or an estimated glomerular filtration rate (eGFR) ≥ 45 mL/min/1.73m2 per Modification of Diet in Renal Disease (MDRD) equation
    * Total serum bilirubin < 2.5 mg/dL (< 5 mg/dL for subjects with known Gilbert's Syndrome)
    * Liver transaminases (AST/ALT/ALP) ≤ 3 × ULN; subjects with liver metastases may have AST, ALT, and ALP ≤ 5 × ULN

Exclusion Criteria:

1. Active CNS metastases, or involvement of the CNS, unless there is a history of at least 3 months of sustained remission of treated disease and no change in steroid dose for at least 28 days prior to study entry.
2. Known past or current malignancy other than inclusion diagnosis, except for:

   1. Cervical carcinoma of stage 1B or less
   2. Noninvasive basal cell or squamous cell skin carcinoma
   3. Noninvasive, superficial bladder cancer
   4. Prostate cancer with a current PSA level < 0.1 ng/mL
   5. Any curable cancer with a CR duration of > 2 years
   6. Enrollment of other malignancies is allowed at the investigator's discretion.
3. Known clinically significant cardiac disease, including:

   1. Onset of unstable angina pectoris within 6 months of signing the informed consent form
   2. Acute myocardial infarction within 6 months of signing the informed consent form
   3. Congestive heart failure (grade II or III or IV as classified by the New York Heart Association)
   4. Impaired cardiac function (LVEF < 50%) as assessed by echocardiogram or MUGA scan
   5. Subjects with uncontrolled arrhythmia or hypertension
   6. Subjects with cardiac valvular disease
4. Unresolved toxicities from prior anticancer therapy, defined as having not resolved per the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) to Grade ≤ 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia, vitiligo, and laboratory test values that otherwise meet inclusion criteria.
5. Ongoing uncontrolled systemic infections requiring antibiotic, anti-fungal, or anti-viral therapy.
6. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, based on laboratory testing performed during screening period. HBV-infected subjects are considered eligible if their viral load is below the institutional limit of quantification (LOQ) and the subject is on stable viral suppressive therapy. HCV infected subjects are considered eligible if they have completed curative antiviral treatment and their HCV RNA viral load is below the institutional LOQ
7. Live vaccine administration planned or required during the treatment period of the trial.
8. History of sensitivity or intolerance to cyclophosphamide or fludarabine.
9. Female subjects of childbearing potential, unable or unwilling to use appropriate contraception (e.g., any combination of condom, diaphragm, intrauterine devices [IUDs], and hormonal oral contraceptives or male partner vasectomy) for the duration of the trial and for 6 months following the last dose of AB-201.

   Male subjects must be sterile (biologically or surgically) or commit to the use of a highly effective method of contraception (any approved combination of physical or chemical methods) until at least 6 months following administration of the last AB-201 dose.)
10. Currently pregnant or lactating (breast feeding must not be started within 6 months of the last dose of AB 201).
11. Any other considerations that might interfere with the assessment of safety or efficacy, or that the investigator deems inappropriate for inclusion.
12. History or presence of a clinically relevant CNS disorder such as seizure disorder (e.g., epilepsy), cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, cerebral edema, posterior reversible encephalopathy syndrome (PRES), or any autoimmune disease with CNS involvement.
13. Any medical, psychological, familial, or sociological conditions that, in the opinion of the Investigator or Sponsor Medical Monitor, would impair the ability of the subject to receive study treatment or comply with study requirements, including understanding and granting informed consent.
14. Severe disease progression or health deterioration within 2 weeks prior to lymphodepletion regimen that, in the opinion of the Investigator, could impair the ability of the subject to receive study treatment or comply with study requirements.
15. Subjects who have undergone organ transplantation
16. Subjects with a history of receiving one or more immune cell therapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Safety & Tolerability (Incidence, severity, seriousness, and dose relationship of Adverse Events) | Up to 18 monthes per patient
  Adverse events and laboratory abnormalities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
Preliminary efficacy, by the objective response rate (ORR) per the Response Evaluation Criteria for Solid Tumors (RECIST) v1.1 | Up to 18 monthes per patient
  The proportion of subjects who experienced an PR or CR, as assessed by investigators per RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- minkyu Jung, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No